CLINICAL TRIAL: NCT05612347
Title: Colonoscopy Versus Stool-based Testing for Older Adults With a History of Colon Polyps
Brief Title: Colonoscopy vs Stool Testing for Older Adults With Colon Polyps
Acronym: COOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Audrey H. Calderwood, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY02001984; PLACER-2020C3-20955 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2022-11-04; First posted 2022-11-10 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Polyp; Colorectal Neoplasms; Colorectal Adenoma; Colorectal Cancer; Digestive System Disease
Keywords: Colonoscopy; Fecal immunochemical test (FIT)
MeSH Terms: conditions — Colorectal Neoplasms; Digestive System Diseases | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FIT (Active Comparator): FIT (annual)
  Interventions: Diagnostic Test: FIT
- Colonoscopy (Active Comparator): Surveillance colonoscopy (one time)
  Interventions: Diagnostic Test: Colonoscopy

INTERVENTIONS:
Diagnostic Test: FIT — Annual FIT
  Arms: FIT
Diagnostic Test: Colonoscopy — One time surveillance colonoscopy
  Arms: Colonoscopy

SUMMARY:
This is a multi-site comparative effectiveness randomized controlled trial (RCT) comparing annual fecal immunochemical testing (FIT) and colonoscopy for post-polypectomy surveillance among adults aged 65-82 with a history of colorectal polyps who are due for surveillance colonoscopy.

DETAILED DESCRIPTION:
Colon polyps are common among adults ≥50 years and people with colon polyps are recommended to undergo regular follow-up colonoscopy (surveillance) in hopes of preventing subsequent colorectal cancer (CRC). Older adults, particularly those who are age ≥70 years, most of whom have a history of only small colon polyps, may benefit little from repeated colonoscopies because of the increased risks of colonoscopy due to age and co-morbidities and potentially limited life expectancy due to other competing medical problems - CRC may never be a problem for them. Older adults may also be hesitant to get repeated colonoscopy because of the risk of complications (e.g., bleeding, perforation, etc.) and inconvenience. More surveillance options are needed to help address the concerns and challenges with repeated colonoscopies in older adults with a history of low-risk polyps.

FIT is a noninvasive, stool-based test that is recommended and widely used in the US and globally for CRC screening in average-risk adults 45 to 75 years of age. In addition, FIT is already standard of care as a surveillance option for patients with a history of low-risk adenomas in Canada and has been shown to be equivalent to colonoscopy for screening of certain high-risk populations (e.g., those with a family history of CRC). However, FIT's role for surveillance among older adults who have a history of low-risk adenomas has not been studied in the US nor among older adults who may benefit from this noninvasive surveillance approach.

The COOP Trial will fill this evidence gap and shed light on patient-, clinician-, and system-factors relevant to FIT for surveillance that together could potentially transform surveillance guidelines in the US and beyond

The purpose of this study is to compare annual at-home stool-based testing, with a fecal immunochemical test (FIT), to colonoscopy in adults age 65-82 who have a history of colorectal polyps. The goal of the study is to compare how well FIT works compared to colonoscopy in looking for and finding colorectal cancer in older adults who have a history of colorectal polyps, as well as to understand people's experiences with using it compared to colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Personal history of colorectal polyps
* Most recent colonoscopy with ≤2 non-advanced polyps
* Currently due or coming due within 12 months for colonoscopy
* Able to provide written informed consent

Exclusion Criteria:

* Personal history of colorectal cancer
* Personal history of genetic syndrome with high risk for colorectal cancer (e.g. Lynch Syndrome, Familial Adenomatous Polyposis Syndrome (FAP), or Serrated Polyposis Syndrome)
* Personal history of inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease)
* Most recent colonoscopy with advanced polyp(s) or ≥3 non-advanced polyps
* Patients unlikely to benefit from polyp surveillance (e.g., history of heart disease or coronary artery disease with treatment in the last 6 months, heart failure affecting function, lung disease requiring use of home oxygen, stroke within the last 4 months, dementia affecting activities of daily living (ADL) or instrumental activities of daily living (IADL), severe liver disease requiring the use of certain medications to control fluid, confusion, or bleeding, severe kidney disease requiring dialysis, or a new cancer diagnosis within the last year)
* Patients unable to provide written informed consent

Ages: 65 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8946 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of advanced neoplasia in each study group, annual FIT and colonoscopy, assessed by comparing the detection of advanced neoplasia between the two study groups. | Up to 11 years
  The investigators will determine the incidence of advanced neoplasia, defined as adenocarcinoma of the colon or rectum or adenomas or serrated polyps ≥1 cm in size or with villous features or any dysplasia, or traditional serrated polyps, in both study groups through annual surveys asking about any changes in polyp history or new cancer diagnosis for up to 6 years and medical record review for up to 11 years. The incidence of advanced neoplasia will be compared between the two study group cumulatively after all the data has been collected.

SECONDARY OUTCOMES:
Change from baseline Satisfaction and Trust of colorectal screening testing assessed by Tiro et al (2005) Response Efficacy sub-scale from the general colorectal cancer screening survey. | Baseline, 1 year after surveillance colonoscopy, annually after each completed FIT for up to 6 years
  The Response Efficacy sub-scale from the general colorectal cancer screening survey is a 2 item scale with five response options (1=strongly disagree, 2=mildly disagree, 3=don't know, 4=mildly agree, 5=strongly agree), such that each individual attains a score ranging from 2 to 10.
Change from baseline worry about colorectal Cancer assessed by the Cancer Worry Scale (CWS) | Baseline and annually for up to 6 years
  The Cancer Worry Scale is a six-item scale designed to measure worry about the risk of developing cancer and the impact of worry on daily functioning. The scale consists of six questions with four response options (1 = not at all or rarely; 2 = sometimes; 3 = often; 4 = almost all the time), such that each individual attains a score ranging from 6 (minimum worry) to 24 (maximum worry).
Change from baseline Perceived colorectal cancer susceptibility using Absolute perceived susceptibility to colorectal polyps subscale from McQueen (2010) | Baseline, annually for up to 6 years
  The absolute perceived susceptibility to colorectal polyps subscale from McQueen (2010) is a three-question scale using four-point Likert format ranging from 1= strongly disagree to 4=strongly agree, such that each individual attains a score ranging from 3 (minimum susceptibility) to 12 (maximum susceptibility).
Change from baseline Emotional benefit of surveillance assessed by a modified version of the Psychological Consequences Questionnaire (PCQ) | Baseline and annually for up to 6 years
  The PCQ is a 22 question scale that has four response options (1=Not at all, 2=a little bit, 3=quite a bit, 4=a great deal) such that each individual attains a score ranging from 22 to 88.
Change from baseline perceived global health assessed by the Patient-Reported Outcomes Measurement Information System-Global 10 | Baseline and annually for up to 6 years
  The Patient-Reported Outcomes Measurement Information System-10 is a 10-item scale that has five response options (5=excellent, 4=very good, 3=good, 2=fair, 1=poor) which assess overall QOL. Raw scores are transformed into T scores; higher T scores indicate greater endorsement of the construct being assessed. Scoring supports two summary scores: A Global Physical Health (GPH) score and a Global Mental Health (GMH) score.
Major and minor harms within 30 days of colonoscopy, as measured through chart review and telephone interview. | 30-45 days post colonoscopy for up to 6 years
  Major and minor harms within 30 days of colonoscopy will be collected through chart review and a telephone interview with participants 30-45 post study surveillance colonoscopy or study colonoscopy for positive FIT. The incidence of harms will be compared between the study groups (annual FIT and colonoscopy).

CONTACTS AND LOCATIONS:
Overall Officials: Audrey H Calderwood, MD, MS, Principal Investigator — Dartmouth-Hitchcock Medical Center; Theodore R Levin, MD, Principal Investigator — Kaiser Permante Northern California
Locations (19):
- United States (17):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Kaiser Permanente Northern California, Walnut Creek, California
  - University of Colorado, Aurora, Colorado
  - MedStar Health, Washington D.C., District of Columbia
  - James A. Haley Veterans Hospital, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Rockford Gastroenterology Associates, Rockford, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, Indiana
  - University of Michigan Health, Ann Arbor, Michigan
  - Dartmouth Health, Lebanon, New Hampshire
  - New York Harbor Health Care System - Dept of Veterans Affairs, New York, New York
  - Kaiser Permanente Northwest, Portand, Oregon
  - Oregon Health & Science University (Knight Cancer Institute), Portland, Oregon
  - Intermountain Health, Sandy City, Utah
  - University of Virginia Health, Charlottesville, Virginia
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta S, Lieberman D, Anderson JC, Burke CA, Dominitz JA, Kaltenbach T, Robertson DJ, Shaukat A, Syngal S, Rex DK. Recommendations for Follow-Up After Colonoscopy and Polypectomy: A Consensus Update by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2020 Mar;158(4):1131-1153.e5. doi: 10.1053/j.gastro.2019.10.026. Epub 2020 Feb 7. No abstract available. PMID 32044092
- [Background] Dubé C, McCurdy BR, Bronstein T, et al. ColonCancerCheck Recommendations for Post-Polypectomy Surveillance, 2019. Available at: https://www.cancercareontario.ca/en/content/coloncancercheck-recommendations-post-polypectomy-surveillance
- [Background] Quintero E, Carrillo M, Gimeno-Garcia AZ, Hernandez-Guerra M, Nicolas-Perez D, Alonso-Abreu I, Diez-Fuentes ML, Abraira V. Equivalency of fecal immunochemical tests and colonoscopy in familial colorectal cancer screening. Gastroenterology. 2014 Nov;147(5):1021-30.e1; quiz e16-7. doi: 10.1053/j.gastro.2014.08.004. Epub 2014 Aug 13. PMID 25127679
- [Background] Kothari ST, Huang RJ, Shaukat A, Agrawal D, Buxbaum JL, Abbas Fehmi SM, Fishman DS, Gurudu SR, Khashab MA, Jamil LH, Jue TL, Law JK, Lee JK, Naveed M, Qumseya BJ, Sawhney MS, Thosani N, Yang J, DeWitt JM, Wani S; ASGE Standards of Practice Committee Chair. ASGE review of adverse events in colonoscopy. Gastrointest Endosc. 2019 Dec;90(6):863-876.e33. doi: 10.1016/j.gie.2019.07.033. Epub 2019 Sep 25. PMID 31563271
- [Background] Warren JL, Klabunde CN, Mariotto AB, Meekins A, Topor M, Brown ML, Ransohoff DF. Adverse events after outpatient colonoscopy in the Medicare population. Ann Intern Med. 2009 Jun 16;150(12):849-57, W152. doi: 10.7326/0003-4819-150-12-200906160-00008. PMID 19528563